CLINICAL TRIAL: NCT05677386
Title: Prevention of Heart Disease in Adult Danes Using Computed Tomography Coronary Angiography - The DANE-HEART Trial
Brief Title: The DANE-HEART Trial - Computed Tomography Coronary Angiography for Primary Prevention
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Herlev Hospital (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Klaus Fuglsang Kofoed, Principle Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DANE-HEART trial
Record Dates: First submitted 2022-12-29; First posted 2023-01-10 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Coronary Atherosclerosis and Other Heart Disease; Cardiovascular Diseases
Keywords: cardiovascular disease; myocardial infarction; CT scans; heart attack
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases; Myocardial Infarction | interventions — Heart Disease Risk Factors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Primary preventive treatment guided by CTCA
  Interventions: Diagnostic Test: Primary preventive treatment guided by CTCA
- Control group (Sham Comparator): Primary preventive treatment guided by Systematic COronary Risk Evaluation (SCORE) 2 model risk assessment according to Danish clinical guidelines.
  Interventions: Other: Cardiovascular risk Score

INTERVENTIONS:
Diagnostic Test: Primary preventive treatment guided by CTCA — Computed tomography coronary angiography (CTCA)
  Other Names: Wide volume CT
  Arms: Intervention group
Other: Cardiovascular risk Score — Systematic COronary Risk Evaluation 2 model for cardiovascular risk prediction
  Other Names: SCORE 2
  Arms: Control group

SUMMARY:
The goal of this randomized controlled clinical trial in asymptomatic individuals with risk factors for cardiovascular disease is to investigate whether a preventive treatment strategy guided by computed tomography coronary angiography (CTCA) provides a patient-centered approach, which ensures optimal protection against serious cardiovascular disease.

The main question it aims to answer is:

Does preventive treatment guided by CTCA reduce the risk of heart attacks or cardiovascular death as compared to using conventional cardiovascular risk scores.

Participants will be randomized to preventive medical therapy and/or invasive intervention guided by either CTCA (intervention group) or Systematic COronary Risk Evaluation (SCORE) 2 model for cardiovascular risk prediction (control group).

DETAILED DESCRIPTION:
The following hypothesis will be tested:

Primary hypothesis: Primary preventive treatment guided by CTCA reduces the risk of myocardial infarction and cardiovascular death compared to standard care in individuals with risk factors for cardiovascular disease.

Additional objectives that will be addressed in the trial include the impact of a CTCA guided preventive treatment strategy compared to standard care with regards to quality of life, adherence to pharmacological preventive therapy, frequency of invasive diagnostic and therapeutic cardiovascular procedures in addition to health economic assessment of cost-effectiveness.

Trial Design

The DANE-HEART Trial is an investigator-initiated, prospective, open label, parallel group, randomized controlled trial assessing the effect of a CTCA guided preventive treatment strategy. Consecutive individuals at risk of cardiovascular disease will be included and randomized 1:1 to the following strategies

Intervention group: Primary preventive treatment guided by CTCA

Control group: Primary preventive treatment guided by Systematic COronary Risk Evaluation (SCORE) 2 risk assessment model according to Danish clinical guidelines.

Patient Cohort

Individuals participating in the Copenhagen General Population Study will be offered participation in the trial. A total of 8000 individuals will be included, or when 6000 individuals have been randomized.

ELIGIBILITY:
Individuals participating in the Copenhagen General Population Study 40 years of age and older, with an estimate glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2 will be offered participation in the trial.

Inclusion Criteria:

Patients must have at least one of the following cardiovascular risk factors:

1. >60 years of age
2. Family history of premature cardiovascular disease (first degree relative with atherosclerotic cardiovascular disease below 60 years)
3. Hypertension (medically treated, or by clinical assessment)
4. Diabetes mellitus
5. Current or recent (within 12 months) smoker
6. Known hypercholesterolaemia (total cholesterol >6.0 mmol/L or receiving statin therapy)
7. Rheumatoid arthritis
8. Systemic lupus erythematosus
9. Chronic kidney disease stage 3 (estimate glomerular filtration rate 30-59 mL/min/1.73 m2).

Exclusion Criteria:

1. CTCA related factors

   * Known persistent atrial fibrillation
   * Known x-ray contrast allergy
   * Implanted intracardiac metal devices
2. Known coronary heart disease or other major atherosclerotic cardiovascular disease

   * Previous coronary revascularization
   * Previous myocardial infarction
   * Heart failure
   * Stroke / Transient ischemic attack
   * Peripheral arterial disease
3. Prior invasive or non-invasive coronary angiography within the last 5 years
4. Known homozygous familial hypercholesterolaemia or other serious inherited disorders of lipid metabolism requiring statin therapy
5. Intolerance of all statins
6. Statin therapy for >2 years

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular death or non-fatal acute myocardial infarction | 5 years
  A composite of cardiovascular death or non-fatal acute myocardial infarction

SECONDARY OUTCOMES:
Acute myocardial infarction | 5 years
  Number of participants with acute myocardial infarction
Heart failure | 5 years
  Number of participants with heart failure
Stroke | 5 years
  Number of participants with stroke
Acute aortic event | 5 years
  Number of participants with acute aortic event
Cardiovascular Events | 5 years
  Number of participants who have fatal and non-fatal myocardial infarction or stroke
Death | 5 years
  Number of all-cause deaths
Coronary cardiovascular procedures | 5 years
  Number of Invasive coronary angiography and coronary revascularisation procedures
Aortic cardiovascular procedures | 5 years
  Number of percutaneous or surgical treatment of aortic disease
Aortic valve procedures | 5 years
  Number of percutaneous or surgical treatments of aortic valve disease
Quality of Life (EQ-5D-5L) | 6 months
  Instrument for Quality of life assessment: Euro Quality of Life - 5 Domain 5 Level (EQ-5D-5L). Value range: 0-100
Quality of Life (EQ-5D-5L) | 2 years
  Instrument for Quality of life assessment: Euro Quality of Life - 5 Domain 5 Level (EQ-5D-5L). Value range: 0-100
Prescriptions | 5 years
  Rates of prescription of preventative therapies
CTCA- incidental findings | Baseline
  Number of participants with incidental findings from CTCA
CTCA related - radiation dose | Baseline
  Radiation dose at baseline CTCA examination

CONTACTS AND LOCATIONS:
Overall Officials: Klaus F Kofoed, MD,SmSc, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Department of Cardiology and Radiology, Rigshospitalet, The Heart Center, Capital Region of Copenhagen, University of Copenhagen, Copenhagen
  - The Copenhagen General Population Study, Herlev-Gentofte Hospital, University of Copenhagen, Denmark, Herlev

IPD SHARING:
Plan to Share IPD: Yes
The intention is to share anonymised data with external collaborators and scientists in according to General Data Protection Regulation rules and Danish laws and regulations.
Supporting Information: Study Protocol, CSR
Time Frame: 1 year after publication of main results
Access Criteria: Requests by email in 2030